CLINICAL TRIAL: NCT03154489
Title: Effectiveness of a Multidisciplinary Medication Review With Follow-up for Patients Treated With Coumarin Anticoagulants in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 914913001
Record Dates: First submitted 2017-04-17; First posted 2017-05-16 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Anticoagulant; Pharmacogenetics; Community Pharmacy Services; Drug Utilization Review; Medication Therapy Management
MeSH Terms: interventions — Acenocoumarol

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acenocoumarol (Other)
  Interventions: Other: acenocoumarol
- control group (Other)
  Interventions: Other: control

INTERVENTIONS:
Other: acenocoumarol — medication review with follow-up in acenocoumarol treatment
  Arms: Acenocoumarol
Other: control — group
  Arms: control group

SUMMARY:
The interdisciplinary collaboration between doctors, nurses and pharmacists, can facilitate the control of patients under treatment with coumarin anticoagulants, increasing their safety and effectiveness. On the other hand, the clinical utility of tools such as pharmacogenetics and the SAME-TT2R2 is unexplored. Based on the foregoing, it seems necessary to study the impact of the Program of medication review with follow-up in collaboration with doctors and nurses in primary care improves the degree of control of the patients under treatment with coumarin anticoagulants. Method: a randomized, controlled study for the main objective. Population and scope of study: Patients on treatment with coumarin anticoagulants with time in therapeutic range (TTR) according to the method of Rosendaal less than 70% in follow-up from primary care in a health area of the Arrabal Health Center (Zaragoza, Spain). Each patient will be followed by a period of 6 months. After this period, patients in the control group (CG) will receive the service of medication review with follow-up for a period of time equivalent (6 months). Intervention: Program of pharmacotherapy follow-up. Variables result: Stability of the INR, drug adherence, intake of vitamin K, knowledge of the patient on the use of acenocoumarol, associated costs, avoided costs, quality of life, satisfaction of patients and professionals involved. Statistical analysis and sample size: 204 patients. Multivariate analysis will be used and cost-effectiveness..

ELIGIBILITY:
Inclusion Criteria:

* Submit a TTR less than 70% in the last 6 months.

Exclusion Criteria:

* Not sign the informed consent.
* Present cognitive difficulties for the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-09-22 (Actual)

PRIMARY OUTCOMES:
Effectiveness of medication review with follow-up | 6 months
  Compare the effectiveness of medication review with follow-up in collaboration with doctors and nurses of primary care patients in treatment with anticoagulants coumarins against the usual practice used actually. Principally studying INR control of this patients during 6 months.

SECONDARY OUTCOMES:
Quality of life related to health | 6 months
  Evaluate the effect of specific pharmaceutical interventions (medication review with follow-up) aimed at patients in treatment with coumarin anticoagulants within the framework of medication review with follow-up quality of life related to health using validated questionnaires.
Study of patients habits | 6 months
  Evaluate the effect of medication review with follow-up on the adherence of the patient, eating habits in relation to the consumption of vitamin K, and their knowledge about the use of acenocoumarol by using validated questionnaires.
Pharmacogenetic analysis of genes CYP2C9 and VKORC1, ApoE CYP4F2 in each patient | 6 months
  Analyze the clinical utility of the incorporation of additional tools like pharmacogenetic analysis of this four genes (CYP2C9 and VKORC1, ApoE CYP4F2) for clinical decision-making in patients with unstable INR. Thanks to the bibliography is known that these gene affect the individual variability of each patient to the acenocoumarol so is going to be studying patients pharmacogenetics for this four genes.
Satisfaction in primary care professionals | 6 months
  Evaluate the satisfaction of medical prescribers, nurses, patients and community pharmacists with the usefulness of medication review with follow-up realized by a pharmacist with focus groups
Review of clinical guidelines used in primary care | 6 months
  Assess therapeutic appropriateness of coumarins anticoagulants in relation to clinical practice guidelines used actually.
Economic outcomes | 6 months
  Evaluate the effect of specific pharmaceutical interventions (medication review with follow-up) aimed at patients in treatment with coumarin anticoagulants within the framework of medication review with follow-up. The economic outcome is going to be assess by following patients if they have admissions in hospital due to bad INR control or they need some extra visits to doctor. This cost a lot to Health System and if it can be avoided it would save costs.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Salud Arrabal, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saez-Benito A, Berenguer N, Magallon R, Olivan B, Ezquerra L, Saez-Benito L. Clinical, economic, and humanistic impact of a multidisciplinary medication review with follow-up for anticoagulated patients treated with vitamin K antagonists in primary care: A cluster randomised controlled trial. Res Social Adm Pharm. 2023 Dec;19(12):1570-1578. doi: 10.1016/j.sapharm.2023.08.007. Epub 2023 Aug 26. PMID 37704534